CLINICAL TRIAL: NCT00546845
Title: Xpert Stent Versus Balloon Angioplasty in Complex Lesions of Small Arteries Below the Knee
Brief Title: Balloon Angioplasty Versus Xpert Stent in CLI Patients XXS Study
Acronym: XXS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Gunnar Tepe MD - University Hospital of Tuebingen, Universtiy hospital of Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XXS
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2007-10

CONDITIONS: Cronic Limb Ishemia; Intervention
MeSH Terms: interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Balloon angioplasty — Balloon angioplasty. Only stent if PTA fails
Device: Use of self-expanding Expert stent — Nitinol stent

SUMMARY:
This study is an investigator-initiated study. The study will be performed as a prospective, randomized, controlled multi-center trial to evaluate the safety and efficiency of Xpert stents compared to PTA in patients with chronic distal artery occlusions or stenosis undergoing catheter revascularization. Patients will be eligible for randomization if they are over 18 years old, if they undergo percutaneous catheter revascularization of an artery below the knee stenosis/occlusion that is less than 15 centimeters in length. Up to two vessels may be treated in this study. All lesions greater than 50% in the below the knee artery region have to be treated either with PTA or stenting according to the randomization.

ELIGIBILITY:
Inclusion Criteria:

Clinical:

1. Age between 18 and 95 years. 2. Subject or subject's legal representative have been informed of the nature of the study, and have signed the patient informed consent form. Patient is willing to take part in the follow-up protocol of the XXS study.

3. Rutherford stage 4 and 5 Anatomical:

1. Additional lesions inflow lesions might be successfully treated before randomization and treatment of the target lesion. The inflow lesions which were treated before randomization should only be classified TASC A or B. (TASC= Trans Atlantic Intersociety Conference)
2. Target vessel with documented run-off to the foot distally of the index lesion with patent plantar arteries
3. Reference vessel diameter of the target lesion should be ≥ 2 and ≤ 5 mm.
4. Maximum treated length in the target vessel is 15 cm (might also be divided up into multiple segments with up to 3 different lesions being treated).
5. Maximum of treated vessels per leg below the knee: 2 (all treated vessels should be treated within the randomization to the study group [PTA or stenting]).
6. Minimum distance target lesion to talus is 5 cm.

Exclusion Criteria:

* Clinical

  1. Life expectancy due to a non-atheroslerotic disease less than 12 months.
  2. Previous bypass surgery < 30 days prior to the study procedure.
  3. Known allergies or sensitivities to heparin, contrast media, aspirin, clopidogrel, and nitinol which cannot be treated with antihistamines.
  4. eGFR less than 29 mL/min/1.73m2 (K-DOQI Class 4 and 5) in patients which are not currently treated with dialysis (equivalent to a serum creatinine level of 2.4 mg/dL in a 70 year old male patient)
  5. Subject with breast feeding plans, or child bearing potential with no birth control.
  6. Subjects enrolled in another study concerning the index vessel(s) within 3 months prior to the study procedure.
  7. Untreatable bleeding diatheses.
  8. Patients who have an indication of being treated with coumadin after the intervention.
  9. Inability to ambulate
  10. Hypercoagulable state
  11. Patients with age <18 years and patients who are not able to sign the informed consent form

Anatomical:

1. Inflow is obstructed and cannot be successfully treated prior to randomization and treatment of below the knee arteries.
2. Acute thrombus present in the target limb.
3. Previously implanted stent in the target vessel(s).
4. Aneurysms in the index leg.
5. Index vessel with no documented run-up to the foot (please also see inclusion criteria, anatomical).
6. Inability to use femoral access
7. No patent pedal arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-09; Primary Completion 2012-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
MLD at the target lesion assessed by angiography | after 12 +/-2 months
  treatment effect dependent if stent of PTA was choosen

SECONDARY OUTCOMES:
1. Interventional success rate. Interventional success is defined as restenosis less than 50%. 2. Late lumen loss (LLL) | after 1, 6, 12 months and 3 years
  treatment effect dependent on the PTA vs. Stent
3. Binary restenosis | arter 6, 12 months and 3 years
  Treament effect in long-term
4. Number of patients initially randomized to the PTA group, but receiving stents because of the suboptimal interventional success. | intervention
  success rate of PTA only
Target lesion revascularization, clinical stage, hospital days | after 1, 6, 12 months, and 3 years
  treatment effect dependet if patients received stents or PTA only

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- Universtiy of Tuebingen, Tübingen, Baden-Wurttemberg, Germany